CLINICAL TRIAL: NCT05322421
Title: Effectiveness of Topical Olive Oil in Prevention and Management of Radiation Induced Oral Mucositis: a Randomised Clinical Control Trial
Brief Title: Effectiveness of Topical Olive Oil in Prevention and Management of Radiation Induced Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salma Hesham Elhoufi (Other)
Responsible Party: Sponsor-Investigator, Salma Hesham Elhoufi, Principal Investiagtor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FDASU-REC 964123
Record Dates: First submitted 2021-11-01; First posted 2022-04-11 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Radiation Mucositis; Oral Mucositis (Ulcerative) Due to Radiation; Radiation-Induced Mucositis
Keywords: radiation; mucositis; oral; stomatitis; olive oil
MeSH Terms: conditions — Stomatitis; Ulcer; Mucositis | interventions — Olive Oil; Sodium Bicarbonate; Solutions

STUDY DESIGN:
Intervention Model Description: This study is designed as a parallel randomized control clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive Oil (Experimental): Will include10 patients receiving topical olive oil application, twice daily
  Interventions: Other: Topical Olive Oil
- Sodium Bicarbonate (Active Comparator): Will include 10 patients receiving Sodium bicarbonate 5% solution, twice daily
  Interventions: Other: Sodium bicarbonate 5% solution

INTERVENTIONS:
Other: Topical Olive Oil — Olive oil will be placed in 200 ml opaque glass containers. For each application, a new stick with a sponge will be submerged into one of the agents to absorb then coat the tongue, buccal mucosa, lips, and hard palate. Patients will be instructed to refrain form eating for 1 hour after the application
  Arms: Olive Oil
Other: Sodium bicarbonate 5% solution — Sodium bicarbonate 5% solution will be placed in 200 ml opaque glass containers. For each application, a new stick with a sponge will be submerged into one of the agents to absorb then coat the tongue, buccal mucosa, lips, and hard palate. Patients will be instructed to refrain form eating for 1 hour after the application
  Arms: Sodium Bicarbonate

SUMMARY:
This research aims to investigate the effectiveness of topical olive oil application both clinically and biochemically as a suitable affordable treatment modality for prevention and management of radiation oral mucositis and its associated pain for head and neck cancer patients receiving radiotherapy.

DETAILED DESCRIPTION:
Twenty adult patients seeking radiotherapy treatment for head and neck cancer are to be selected. Patients meeting the eligibility criteria are to be equally and randomly allocated in 2 different groups. Group 1 will include10 patients receiving topical olive oil application, twice daily (Experimental arm). Group 2 will include 10 patients receiving Sodium bicarbonate 5% solution, twice daily (Control arm). Both intervention and control groups will start the application of the agents two days before the induction of radiotherapy. Evaluation will be done using World Health Organization (WHO) scale for oral mucositis to record the extent and severity of oral mucositis. Pain and discomfort will be evaluated using Numeric Rating Scale (NRS). Clinical evaluation using both scales will be performed after starting radiotherapy every other week ( after 2 weeks, after 4 weeks and after 6 weeks at the end of the treatment). Patients scores will be recorded at similar intervals. Total Antioxidant Capacity "TAC" will be used to study the biochemical effect of topical olive oil application by evaluating the oxidative stress in the saliva. Saliva samples will be collected from all patients of both groups prior to the beginning of radiotherapy, and a second sample will be collected after six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged above 25 years up to 65 years.
* Both genders are eligible.
* Patients with head and neck cancer who are planned to receive radiotherapy either as postoperative (adjuvant after surgery) or definitive therapy.
* Patients planned to receive radiotherapy treatment with a dose of 60-70 Gy.

Exclusion Criteria:

* Patients with known sensitivity to olive oil and/or any of its products
* Patients with gingival or oral ulceration or mucositis
* Smokers
* Vulnerable patients (pregnant women, neonates, children, prisoners, persons with physical handicaps or mental disabilities)
* Pregnant and lactating women.
* Patients with any uncontrolled systemic diseases (such as diabetes, cardiovascular, liver disorder, renal dysfunction)
* Patients suffering from any physical or mental disabilities that would interfere with or be affected by the study procedure.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Oral Radiation mucositis | Every other week ( 2 weeks, 4 weeks and 6 at the end of the treatment)
  Number of participants who develop Radiation mucositis according to the WHO Scale. (grade 0 indicates that no changes have occurred in the oral cavity and grade 4 indicates the worst level of mucositis )
Grade of oral radiation mucositis | Every other week ( 2 weeks, 4 weeks and 6 weeks at the end of the treatment)
  Clinical evaluation using the WHO scale will be performed to record the changes in the oral cavity after starting radiotherapy, (grade 0 indicates that no changes have occurred in the oral cavity and grade 4 indicates the worst level of mucositis )

SECONDARY OUTCOMES:
Post operative pain assessment using Numeric Pain Rating Scale | Patients scores will be recorded after starting radiotherapy every other week ( 2 weeks, 4 weeks and 6 weeks at the end of the treatment)
  To evaluate patient's perception of postoperative pain during the treatment time using the NRS (Numeric Pain Rating Scale). The NRS is an 11-point numeric scale that ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Total antioxidant capacity | Salivary samples will be collected at baseline before the induction of radiotherapy and at 6 weeks at the end of the treatment for TAC analysis.
  To evaluate the biochemical effect of topical olive oil application using the Total Antioxidant Capacity (TAC) test in the saliva of patients with radiation oral mucositis

CONTACTS AND LOCATIONS:
Overall Officials: Suzan S Ibrahim, Professor, Study Director — Ain Shams University; Radwa Ragheb, Lecturer, Study Director — Ain Shams University; Salma H Elhoufi, Principal Investigator — Ain Shams University
Locations (1):
- Salma Hesham Elhoufi, Cairo, Select, Egypt

IPD SHARING:
Plan to Share IPD: No